CLINICAL TRIAL: NCT01713452
Title: A Randomized Trial of Ostomy Closure Techniques: An Outcomes Evaluation of Primary Closure Versus Pursestring Closure
Brief Title: A Randomized Trial of Ostomy Closure Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0806M37362
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Wound Infection
Keywords: Surgical Stomas; ileostomy; surgical site infection
MeSH Terms: conditions — Wound Infection; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purse string closure (Active Comparator): Patients undergo a purse string closure of their old stoma site.
  Interventions: Procedure: Purse string closure
- Primary closure (Active Comparator): Patients have their stoma sites close primarily with staples.
  Interventions: Procedure: Primary closure

INTERVENTIONS:
Procedure: Purse string closure — 1. An incision around the stoma will be made with 2-3 mm circumferential margins. This dissection along the mucocutaneous junction will then be made to the fascial defect. Re-establishment of bowel continuity will them be performed. If the circumferential incision does not provide adequate exposure, the incision can be converted to an elliptical one. Thereafter, it will be closed primarily with staples, similar to the primary closure group.
  2. Following ostomy closure, the subcutaneous tissues will be irrigated. A 2-0 monocryl subcuticular purse string stitch will then be placed and cinched to a 1cm diameter. This opening will then be packed with Nu-Gauze as a wick dressing.
  3. Diameter of the skin defect should then be measured.
  4. A postoperative photo will then be taken.
  Arms: Purse string closure
Procedure: Primary closure — 1. An elliptical incision (extending transversely) will be made with 2-3 mm superior/inferior margins around the mucocutaneous junction. Dissection will then be made in a perpendicular fashion through the subcutaneous tissue with tapering near the fascial defect. Re-establishment of bowel continuity will then be performed.
  2. Following ostomy closure, the subcutaneous tissue will be irrigated and the skin will be closed tight with staples placed at close intervals (<1.5cm). No subcutaneous drains will be placed.
  3. Length of the incision should be measured in centimeters.
  4. A postoperative photo will then be taken.
  Arms: Primary closure

SUMMARY:
Stoma closure has been associated with a high rate of surgical site infection (SSI). The rate for SSI following stoma closure has been noted to be 7-41%; a rate that is higher than expected for a clean-contaminated operative classification. The ideal stoma site closure technique is still debated in the current literature. The aim of this study was to compare the rate of SSI following two different stoma closure techniques, primary closure versus a skin approximating purse string closure, in a multi-center randomized controlled trial. The investigators hypothesize that purse string closure technique will have a lower rate of SSI than primary closure technique.

DETAILED DESCRIPTION:
The investigators will randomize ileostomy takedown patients to either a primary closure or purse string closure technique intraoperatively. Surgeons at both the University of Minnesota and the CHUV hospital in Switzerland will participate in the this study.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible are those with either a colostomy or ileostomy (end or loop) who are deemed by their surgeon to be appropriate candidates for ostomy closure. There will be no limitations based upon initial indication for formation of the ostomy. Indications for initial ostomy formation for fecal diversion can include: infection (e.g. diverticulitis) and protection of an anastomosis. (following resection for inflammatory bowel disease, benign diseases, or cancer)

Exclusion Criteria:

Subjects will be excluded from the study if:

1. The stoma site is left open to heal by secondary intention due to gross contamination (surgeon discretion)
2. The stoma site is re-used (i.e. the same stoma site used for the formation of a new ostomy)
3. A new stoma is created at a different site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-12; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
surgical site infection | 30 days postoperatively

SECONDARY OUTCOMES:
delayed wound healing | 30 days postoperatively
  Evidence of delayed wound-healing at stoma takedown site
patient satisfaction | 30 days postoperatively
  We are measuring subject satisfaction with wound healing and cosmetic outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Lee JT, Marquez TT, Clerc D, Gie O, Demartines N, Madoff RD, Rothenberger DA, Christoforidis D. Pursestring closure of the stoma site leads to fewer wound infections: results from a multicenter randomized controlled trial. Dis Colon Rectum. 2014 Nov;57(11):1282-9. doi: 10.1097/DCR.0000000000000209. PMID 25285695